CLINICAL TRIAL: NCT01039844
Title: Phase I Study of Weekly LOC-paclitaxel Injection
Brief Title: Study of Weekly LOC-paclitaxel Injection for Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0432; NCI-2011-01188 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Melanoma
Keywords: LOC-paclitaxel Injection; metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Weekly LOC-paclitaxel Injection (Experimental): LOC-paclitaxel IV by a 1 hour infusion on Day 1, 8, 15, 22 and 29; repeated every 42 days (6 weeks) per cycle.
  Interventions: Drug: LOC-paclitaxel

INTERVENTIONS:
Drug: LOC-paclitaxel — Phase I Starting Dose: 100 mg/m^2 IV (intravenously) 1 hour infusion on Day 1, 8, 15, 22 and 29; and repeated every 42 days (6 weeks) per cycle.
  Phase II Starting Dose: Maximum tolerated dose from Phase I.

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of LOC-paclitaxel when given to patients with metastatic melanoma. The safety of this drug and if it can control the disease is also being studied.

DETAILED DESCRIPTION:
The Study Drug:

Paclitaxel is designed to block cancer cells from dividing, which may cause them to die. LOC-paclitaxel is a redesigned version of paclitaxel. Fatty acid is added to paclitaxel, which may help paclitaxel to stay in the tumor for longer at higher concentrations. This is the first study using LOC-paclitaxel in humans.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of LOC-paclitaxel based on when you joined this study. Up to 9 dose levels of LOC-paclitaxel will be tested. Three (3) to 6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of LOC-paclitaxel is found.

Once the highest tolerable dose of LOC-paclitaxel is found, 12 participants will receive the study drug at that dose level.

Study Drug Administration:

Each study cycle is 6 weeks.

You will receive LOC-paclitaxel by vein over 1 hour on Days 1, 8, 15, 22, and 29 of each cycle.

If you experience side effects, your dose of study drug may be lowered.

Study Visits:

On Day 1 of each cycle:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 1 tablespoon) will be drawn for routine tests and to test for tumor markers.
* If you have melanoma of the head and neck, you will have a CT scan of the neck.
* If you have skin lesions, photographs will be taken of the lesions. Your private areas will be covered (as much as possible), and a picture of your face will not be taken unless there are lesions on your face. You will not be able to be identified by any pictures that may be taken of your lesions.

Once a week:

* Blood (about 1 teaspoon) will be drawn to check your blood cell counts.
* Urine will be collected for routine tests.
* You will be asked if you experienced any side effects.

Every 6 weeks, you will have x-rays and CT scans to check the status of the disease as per standard of care. If you have had a response to treatment (the disease has disappeared or the tumors have gotten smaller), the x-rays and CT scans will be repeated again in 4 weeks. After that, they will be repeated every 6 weeks.

If you experience low blood counts while you are on study, and the doctor thinks it is severe, you will have a bone marrow biopsy to check for the cause of the low blood counts.To collect a bone marrow biopsy, an area of the hip is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle.

If the doctor thinks it is needed, you will have ECGs and extra blood (about 1 teaspoon) will be drawn.

Any of the procedures listed in this consent form may be performed more frequently, if your doctor thinks they are needed.

Pharmacokinetic (PK) Testing:

Extra blood will also be drawn for PK testing. PK testing measures the amount of study drug in the body at different time points. Blood (about 2 teaspoons each time) will be drawn at the following times:

* On Day 1 of Cycle 1, blood will be drawn before the dose of LOC-paclitaxel, at the end of the dose, and then 5 more times over the next 11 hours after the dose.
* On Days 2-7 of Cycle 1, blood will be drawn 1 time each day.
* On Days 8, 15, and 22 of Cycle 1, blood will be drawn 1 time each day.
* On Day 29 of Cycle 1, blood will be drawn before the dose, at the end of the dose, and then 5 more times over the next 11 hours after the dose.
* On Days 30-35 of Cycle 1, blood will be drawn 1 time each day.

Length of Study:

You will be on study for as long as you are benefiting. You will be taken off the study if you experience intolerable side effects or the disease gets worse.

End-of-Study Visit:

After you are off study, you will have an end-of-study visit. At this visit, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 1 tablespoon) will be drawn for routine tests and to measure tumor markers.
* You will have CT scans to check the status of the disease.
* If you are having low blood counts, you will have a bone marrow biopsy to check for side effects.
* If you have skin lesions, photographs will be taken of the lesions.

After you go off study, extra tests may be needed for your safety. This may include routine blood tests (about 1 tablespoon) and will be continued until you have recovered from any side effects, which may be 3-4 weeks.

This is an investigational study. LOC-paclitaxel is not FDA approved or commercially available. LOC-paclitaxel is currently being used for research purposes only.

Up to 60 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have histologically or cytologically confirmed malignant solid tumors.
2. Patients must have failed conventional therapy for their cancer or have a malignancy for which a conventional therapy does not exist.
3. Patients must have recovered from all acute toxicities from prior therapies, excluding alopecia.
4. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
5. Patients must be >/= 18 years of age.
6. Patients must have adequate liver and renal function as defined by serum creatinine, total bilirubin, AST, and ALT levels within normal limits.
7. Patients must have adequate bone marrow function as defined by a hemoglobin >/= 10g/dL, an absolute neutrophil count of >/= 1,500/mm^3, and platelet count of >/= 100,000/mm^3.
8. Patients must sign an informed consent form indicating that they are aware of the investigational nature of this study and in keeping with the policies of the institution.
9. Patients must have a life expectancy of at least three months.

Exclusion Criteria:

1. Patients who have therapies available that have demonstrated clinical benefit.
2. Patients with known or clinical evidence of central nervous system (CNS) metastases.
3. Women who are pregnant or nursing and patients (men or women) who are not practicing an acceptable method of birth control. A negative pregnancy test (urine or serum) must be documented at baseline for women of childbearing potential. Women may not breastfeed while on this study.
4. Patients with current active infections requiring anti-infectious treatment (e.g., antibiotics, antivirals, or antifungals).
5. Patients with current peripheral neuropathy of any etiology that is greater than grade 1.
6. Patients with unstable or serious concurrent medical conditions are excluded. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent.
7. Patients with a known hypersensitivity to CREMOPHOR® and/or paclitaxel.
8. Patients must not have had recent major surgery within the past 14 days or large field radiation therapy or chemotherapy in the last 28 days. If the previous chemotherapy included nitrosoureas or mitomycin C, this period will be 6 weeks.
9. Patients must not receive any concurrent chemotherapy, radiotherapy, or immunotherapy while on study. Previous palliative radiotherapy is allowed for metastatic disease in a region that is not part of the disease being measured.
10. Patients must not have had radiation to >/= 25% of the bone marrow.
11. Patients with Gilbert's Syndrome.
12. Patients with known HIV disease or infection.
13. Simultaneous participation in another clinical trial of an investigational agent or device.
14. Patients receiving ketoconazole, erythromycin, verapamil, diazepam, quinidine, diltiazem, rifampicin, carbamazepine, phenytoin, efavirenz, nevirapine, fluoxetine or gemfibrozil. Patients taking any of these drugs may qualify for treatment on this investigational study if they have been off the drug at least for 7 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of LOC-Paclitaxel | 6 week cycles
  MTD defined as the dose of LOC-paclitaxel at which no more than 2 of 6 patients experience dose limiting toxicity (DLT).
Toxicity of Weekly LOC-Paclitaxel | Day 1 of each 6 week cycle
  Toxicity will be graded according to the NCI Common Toxicity Criteria (CTC), Version 3.0.
Tumor Response | 6 weeks
  The Response Evaluation Criteria in Solid Tumors (RECIST) used to assess tumor response to treatment in this study. Complete Response (CR): disappearance of all target lesions determined by two consecutive observations not less than four weeks apart. Partial Response (PR): at least a 30% decrease in the sum of longest diameter (LD) of target lesions taking as reference the baseline sum LD determined by two consecutive observations not less than four weeks apart.
  Progression (PD): at least a 20% increase in the sum of LD of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD since the treatment started.

CONTACTS AND LOCATIONS:
Overall Officials: Rodabe N. Amaria, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org